CLINICAL TRIAL: NCT04564469
Title: Influence of Diuresis Timing (F+0 Vs F-15) on 99m Tc DTPA Renography for the Diagnosis of Suspected Obstructive Uropathy in Adult Hydronephrotic Patients.
Brief Title: Influence of Diuresis Timing (F+0 Vs F-15) on 99m Tc DTPA Renography for the Diagnosis of Suspected Obstructive Uropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Gamal Fathy, Resident doctor, Assiut University
Other Study IDs: F+0 Vs F-15 in renal scan
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Renal Scan in Suspected Obstructive Uropathy in Adult Hydronephrotic Patient
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Furosemide — A number of different protocols exist in terms of the timing of furosemide injection, (F+0) protocol in which furosemide is injected at the same time of radiotracer administration &( F - 15)protocol in which furosemide is administered 15 min before tracer administration

SUMMARY:
Evaluation of the influence of the diuretic injection timing (F+0 Vs F-15) on the dynamic 99mTc- DTPA renal scintigraphy for the diagnosis of suspected obstructive uropathy in adult hydronephrotic patients.

DETAILED DESCRIPTION:
Obstructive uropathy can be defined as any blockage of urine drainage from the kidney (renal calyces or renal pelvis), ureter, or bladder. As a result of the blockage, urine backs up into the kidneys, causing dilatation of the ureter, renal pelvis, and renal calyces, which can damage the kidney if it is not treated. The appearance of dilated or enlarged renal pelvis and calyces is referred to as hydronephrosis and is a symptom of obstructive uropathy.

Diuresis renography(renal scan with using of diuretic drug such as furosemide) is non-invasive test which is based on a high endogenous rate of urine flow stimulated by the administration of furosemide. Interpretation of the test is based on the rate of washout of the radiopharmaceutical from the collecting system in the upper urinary tract.

A number of different protocols exist in terms of the timing of furosemide injection, (F+0) protocol in which furosemide is injected at the same time of radiotracer administration &( F - 15)protocol in which furosemide is administered 15 min before tracer administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years.
* Patients with hydronephrosis (unilateral or bilateral) referred for renal scan.
* Patients able to sleep in a fixed position for 20 minutes.

Exclusion Criteria:

* Severely impaired renal function.
* Advanced hydronephrosis
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patient equal to or more than 18 years old with hydronephrosis and able to be stable on table for 20 minutes not pregnant ,not presented with severe renal impairement&not presented with severe hydronephrosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Comparison between F+0 and F-15 diuretic protocols to differentiate between functional renal obstruction from mechanical obstruction in adult hydronephrotic patients. | One year
  Analysis of T1/2 in renal scan and find which time of furosemide injection give conclusive results in dignosis of obstructive uropathy

REFERENCES:
- [Background] Taylor AT, Brandon DC, de Palma D, Blaufox MD, Durand E, Erbas B, Grant SF, Hilson AJW, Morsing A. SNMMI Procedure Standard/EANM Practice Guideline for Diuretic Renal Scintigraphy in Adults With Suspected Upper Urinary Tract Obstruction 1.0. Semin Nucl Med. 2018 Jul;48(4):377-390. doi: 10.1053/j.semnuclmed.2018.02.010. Epub 2018 Mar 16. No abstract available. PMID 29852947
- [Background] Gordon I, Piepsz A, Sixt R; Auspices of Paediatric Committee of European Association of Nuclear Medicine. Guidelines for standard and diuretic renogram in children. Eur J Nucl Med Mol Imaging. 2011 Jun;38(6):1175-88. doi: 10.1007/s00259-011-1811-3. PMID 21503762